CLINICAL TRIAL: NCT01630863
Title: The Safe Effective Light Dose of Photodynamic Therapy for Chronic Central Serous Chorioretinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Min Sagong, Assistant Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YUH-12-007-D4
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Central serous chorioretinopathy; photodynamic therapy; safe and effective dose
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Photochemotherapy

ARMS (3):
- 50% group (Experimental): power of PDT is applied to the patients at 50% of the full energy based on TAP study.
  Interventions: Procedure: Photodynamic therapy
- 40% group (Experimental): Decreasing power of PDT is applied to the patients at 40% of the full energy based on TAP study.
  Interventions: Procedure: Photodynamic therapy
- 30% group (Experimental): Decreasing power of PDT is applied to the patients at 30% of the full energy based on TAP study.
  Interventions: Procedure: Photodynamic therapy

INTERVENTIONS:
Procedure: Photodynamic therapy — Photodynamic therapy is performed using verteporfin. Full dose of verteporfin is infused for 10 minutes, followed by laser delivery at 15 minutes from the start of infusion. Different light dose of PDT is applied to the patients at 50%, 40% and 30% of the full energy based on TAP study. The area of irradiation is set to the abnormal choroidal vascular hyperpermeability on ICGA corresponding to the leaking area on FA.

SUMMARY:
To find the safe effective lowest light dose for photodynamic therapy (PDT). in the treatment of central serous chorioretinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic detachment of the neurosensory retina with a focal leak at the level of the RPE with FA
2. Presence of SRF and/or serous pigment epithelial detachment on optical coherence tomography (OCT)
3. Presence of abnormal dilated choroidal vasculature in ICGA
4. Patients with symptomatic CSC of at least 3 months duration

Exclusion Criteria:

1. Patients who received any previous treatment, including PDT or focal thermal laser photocoagulation for CSC, or who had evidence of CNV, PCV, or other maculopathy on clinical examination, FA, or ICGA
2. Patients receiving exogenous corticosteroid treatment
3. Patients with systemic diseases such as Cushing's disease or renal diseases
4. Pregnant patients

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Changes of best corrected visual acuity | 6 month
  Changes of best corrected visual acuity at baseline and 1, 3, 6 month after PDT

SECONDARY OUTCOMES:
Change of central retinal thickness, success rate, recurrence rate, and complications | 6 months
  Change of the central retinal thickness on optical coherence tomography (OCT)are compared at baseline at 1, 3, and 6 months after PDT. Additionally, success rate, recurrence rate, and complications between three groups are evaluated during 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University College of Medicine, Daegu, South Korea

REFERENCES:
- [Derived] Park DG, Jeong S, Noh D, Sagong M. Optimal fluence rate of photodynamic therapy for chronic central serous chorioretinopathy. Br J Ophthalmol. 2021 Jun;105(6):844-849. doi: 10.1136/bjophthalmol-2020-316837. Epub 2020 Jul 29. PMID 32727733